CLINICAL TRIAL: NCT04630028
Title: A Phase 3 Study of the Efficacy, Safety and Pharmacokinetics of Ustekinumab as Open-label Intravenous Induction Treatment Followed by Randomized Double-blind Subcutaneous Ustekinumab Maintenance in Pediatric Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Ustekinumab in Pediatric Participants With Moderately to Severely Active Ulcerative Colitis (UC)
Acronym: UNIFI Jr
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108865; CNTO1275PUC3001 (Other: Janssen Research & Development, LLC); 2019-004224-38 (EudraCT Number); 2023-504977-19-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Weights and Measures; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Induction Period (I): Ustekinumab (Experimental): All participants will receive a single intravenous (IV) administration of ustekinumab at induction Week 0 (I-0) based on body surface area (BSA) (milligram per meter square [mg/m^2]) or weight-tiered induction dose (milligram per kilogram [mg/kg]).
  Interventions: Drug: Ustekinumab Dose Based on BSA and Body Weight
- Maintenance (M) Period: Ustekinumab once every 8 Week (q8w) (Experimental): Participants will receive subcutaneous (SC) administration of ustekinumab every 8 weeks (q8w) based on BSA (mg/m^2) or weight-tiered induction dose (mg/kg) at Weeks M-0, M-8, M-16, M-24, M-32, M-40 and matching placebo at Weeks M-12 and M-36 to maintain the blind.
  Interventions: Drug: Ustekinumab Dose Based on BSA and Body Weight; Drug: Matching Placebo
- Maintenance (M) Period: Ustekinumab once every 12 Week (q12w) (Experimental): Participants will receive SC administration of ustekinumab every 12 weeks (q12w) based on BSA (mg/m^2) or weight-tiered induction dose (mg/kg) at Weeks M-0, M-12, M-24, M-36 and matching placebo at Weeks M-8, M-16, M-32, and M-40 to maintain the blind.
  Interventions: Drug: Ustekinumab Dose Based on BSA and Body Weight; Drug: Matching Placebo

INTERVENTIONS:
Drug: Ustekinumab Dose Based on BSA and Body Weight — As per BSA and body weight Ustekinumab will be administered SC and IV.
  Other Names: STELARA
Drug: Matching Placebo — Placebo will be administered subcutaneously.
  Arms: Maintenance (M) Period: Ustekinumab once every 12 Week (q12w); Maintenance (M) Period: Ustekinumab once every 8 Week (q8w)

SUMMARY:
The purpose of this study is to evaluate: a) the efficacy of ustekinumab dosing in inducing clinical remission, b) safety profile of ustekinumab, and c) ustekinumab exposure (pharmacokinetics [PK]) in pediatric participants with moderately to severely active UC.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable on the basis of physical examination, medical history, and vital signs, performed at screening. Any abnormalities must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and acknowledged by the investigator
* Must have had UC diagnosed prior to screening
* Have moderately to severely active UC, defined as a baseline Mayo score of 6 through 12, inclusive, with a screening Mayo endoscopy subscore greater than or equal to (>=) 2 as determined by a central review of the video of the endoscopy
* A participant who has had extensive colitis for >= 8 years, or disease limited to the left side of the colon for >= 10 years, must: a) have had a full colonoscopy to assess for the presence of dysplasia within 1 year before the first administration of study intervention or b) have a full colonoscopy with surveillance for dysplasia as the baseline endoscopy during the screening period. Results from these surveillance biopsies must be negative for dysplasia (low-grade, high-grade, or indeterminant) prior to the first administration of study intervention
* Females of childbearing potential must have a negative highly sensitive urine pregnancy test at screening and at Week I-0 prior to study intervention administration

Exclusion Criteria:

* Have UC limited to the rectum only or to less than (<) 20 centimeter (cm) of the colon
* Presence or history of colonic or small bowel obstruction within 6 months prior to screening, confirmed by objective radiographic or endoscopic evidence of a stricture with resulting obstruction (dilation of the colon or small bowel proximal to the stricture on barium radiograph or an inability to traverse the stricture at endoscopy)
* Have a history of latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis, or have had a nontuberculous mycobacterial infection prior to screening
* Presence or history of any malignancy including presence or history of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (example, nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic areas) and monoclonal gammopathy of undetermined significance, or clinically significant hepatomegaly or splenomegaly
* Has known allergies, hypersensitivity, or intolerance to ustekinumab or its excipients

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Global: Number of Participants with Clinical Remission at Induction Week 8 (I-8) Visit | Week 8
  Clinical remission is defined as Mayo stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 74 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability | Up to 74 weeks
  SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, and suspects transmission of any infectious agent via a medicinal product.
Number of Participants with AEs Leading to Discontinuation of Study Intervention | Up to 74 weeks
  Number of Participants with discontinuation of study intervention due to an AE, infections, injection-site reactions, and AEs during or within 1 hour of an infusion will be reported.
Number of Participants with AEs of Special Interest (AESI) as a Measure of Safety and Tolerability | Up to 74 weeks
  AESI of any newly identified malignancy, case of active tuberculosis (TB), or opportunistic infection occurring after the first administration of study intervention(s) in participants will be reported.
Number of Participants with Laboratory Abnormalities | Up to 74 weeks
  Number of participants with laboratory abnormalities related to hematology, serum chemistry, and coagulation will be reported.
Reactions Temporally Associated with an Intravenous (IV) Infusion and Subcutaneous (SC) Injection-site Reactions | Up to 74 weeks
  Reactions temporally associated with an IV infusion (induction period) and SC injection-site reactions (maintenance period) will be reported.
Serum Concentration of Ustekinumab | Up to 74 weeks
  Serum samples will be analyzed to determine concentrations of ustekinumab.
US Specific: Clinical Remission at M-44 for Participants who are in Clinical Response at I-8 | Week 52
  Clinical remission at M-44 for participants who are in clinical response at I-8 will be reported. Clinical remission is defined as a Mayo stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline.

SECONDARY OUTCOMES:
Number of Participants With Clinical Response at I-8 Visit | Week 8
  Clinical response is defined as decrease from baseline in the modified Mayo score by >= 30 percent (%) and >=2 points, with either a decrease from baseline in the rectal bleeding subscore of >= 1 or a rectal bleeding subscore of 0 or 1.
Number of Participants with Symptomatic Remission at I-8 Visit | Week 8
  Symptomatic remission is defined as Mayo stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0, where the stool frequency subscore has not increased from induction baseline.
Clinical Remission at I-8 as Assessed by the Pediatric Ulcerative Colitis Activity Index Score (PUCAI) Score | Week 8
  Clinical remission is defined as a PUCAI score less than (<)10.
Endoscopic Improvement at I-8 Visit | Week 8
  Endoscopic improvement is defined as a Mayo endoscopy subscore of 0 or <= 1 with no friability present on the endoscopy.
Histologic-endoscopic Mucosal Improvement at Week I-8 | Week 8
  Histologic-endoscopic mucosal improvement is defined as achieving a combination of histologic (neutrophil infiltration in less than [<] 5% of crypts, no crypt destruction, and no erosions, ulcerations or granulation tissue according to the Geboes grading system) and endoscopic improvement (endoscopy subscore of 0 or 1 with no friability present on the endoscopy).
Number of Participants with Clinical Remission at Week 44 (M-44) Visit | Week 52
  Clinical remission is defined as a Mayo stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline.
Number of Participants with Symptomatic Remission at M-44 Visit | Week 52
  Symptomatic remission is defined as Mayo stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0, where the stool frequency subscore has not increased from induction baseline.
Clinical Remission at M-44 as Assessed by the PUCAI Score | Week 52
  Clinical remission is defined as a PUCAI score less than < 10.
Endoscopic Improvement at M-44 Visit | Week 52
  Endoscopic improvement is defined as a Mayo endoscopy subscore of 0 or <= 1 with no friability present on the endoscopy.
Corticosteroid-free Clinical Remission at Week M-44 | Week 52
  Corticosteroid-free clinical remission is defined as a Mayo stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline; and not receiving corticosteroids for at least 90 days prior to Week M-44.
Clinical Remission at M-44 and not Receiving Corticosteroids for at Least 90 Days Prior to M-44 Among Participants who Received Corticosteroids at M-0 | Week 52
  Clinical remission is defined as a PUCAI score less than < 10. Clinical remission at M-44 and in participants not receiving corticosteroids for at least 90 days prior to M-44 among participants who received corticosteroids at M-0 as assessed by PUCAI score will be reported.
Clinical Remission at M-44 for Participants who are in Clinical Remission at I-8 | Week 52
  Clinical remission at M-44 for participants who are in clinical remission at I-8 will be reported. Clinical remission is defined as a Mayo stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline.
US Specific: Number of Participants with Clinical Remission at I-8 Visit | Week 8
  Clinical remission is defined as Mayo stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline.
Histologic-endoscopic Mucosal Improvement at Week M-44 | Week 52
  Histologic-endoscopic mucosal improvement is defined as achieving a combination of histologic (neutrophil infiltration in < 5% of crypts, no crypt destruction, and no erosions, ulcerations or granulation tissue according to the Geboes grading system) and endoscopic improvement (endoscopy subscore of 0 or 1 with no friability present on the endoscopy).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (58):
- United States (9):
  - Nemours DuPont Hospital for Children, Wilmington, Delaware
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Levine Childrens at Atrium Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Cook Childrens Medical Center, Fort Worth, Texas
  - Pediatric Specialists Of Virginia, Fairfax, Virginia
- Belgium (5):
  - Universitair Kinderziekenhuis Koningin Fabiola, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Gent, Ghent
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
- Germany (8):
  - Universitätsklinikum Aachen, Aachen
  - Charite-Universitätsmedizin Berlin - Berlin, Berlin
  - Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Dr. von Haunersches Kinderspital, Munich
  - KUNO Klinik St. Hedwig, Regensburg
  - Universitatsklinikum Ulm, Ulm
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod Abauj Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szabolcs Szatmar Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - Szegedi Tudományegyetem, Gyermekgyógyászati Klinika és Gyermekegészségügyi Centrum, Szeged
- Israel (6):
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Japan (9):
  - Juntendo University Hospital, Bunkyō City
  - Gunma University Hospital, Gunma
  - Kindai University Nara Hospital, Ikoma
  - Kurume University Hospital, Kurume
  - Saitama Childrens Medical Center, Saitama Shi
  - Miyagi Children's Hospital, Sendai
  - National Center for Child Health and Development, Setagaya Ku
  - Jichi Medical University Hospital, Shimotsuke
  - Mie University Hospital, Tsu
- Poland (6):
  - Szpital im. M. Kopernika, Gdansk
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - GASTROMED Sp. z o.o., Torun
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Russia (6):
  - Kazan State Medical University, Kazan'
  - Russian National Research Medical University named after N.I.Pirogov, Moscow
  - FSBI 'Scientific Centre of Children Health' of the Russian Academy of Medical Sciences, Moscow
  - Privolzhsky Research Medical University of Ministry of Health of Russian Federation, Nizhny Novgorod
  - Saratov State Medical University, Saratov
  - Yaroslavl Regional Children's Clinical Hospital, Yaroslavl
- United Kingdom (4):
  - Birmingham Children's Hospital, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency